CLINICAL TRIAL: NCT00396890
Title: Enhancing Interhemispheric Disinhibition Between Motor Cortices Using Bilateral Brain Stimulation
Brief Title: Enhancing Brain Activity With Magnetic Stimulation
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070022; 07-N-0022
Record Dates: First submitted 2006-11-07; First posted 2006-11-08 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-12-15

CONDITIONS: Healthy
Keywords: Theta Burst Stimulation; Repetitive TMS (rTMS); Transcranial Magnetic Stimulation (TMS); Primary Motor Cortex; Interhemispheric Disinhibition; Healthy Volunteer; HV

SUMMARY:
This study will determine whether stimulation of the right side of the brain with repetitive transcranial magnetic stimulation (rTMS) followed by stimulation of the left side with theta burst stimulation (TBS) can temporarily change brain activity and improve hand movements in subjects more than has recently been achieved with rTMS alone.

For rTMS, a wire coil is held on the patient's scalp. A brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. The subject hears a click and may feel a pulling sensation on the skin under the coil. There may be a twitch in the muscles of the face, arm or leg. The subject may be asked to tense certain muscles slightly or perform other simple actions. The effect of TMS on the muscles is detected with small metal disk electrodes taped to the skin of the arms or legs. This study uses two kinds of rTMS. In one (Hz rTMS), magnetic pulses are given once per second for a period of 20 minutes; in the other (TBS), a series of pulses are given in bursts, each lasting 2 seconds, for a period of 3 minutes.

Healthy normal volunteers between 18 and 55 years of age may be eligible for this study. Participants undergo the following procedures during three visits to the NIH Clinical Center:

Visit 1:

Participants receive either real or sham rTMS applied on the right side of the brain followed by real or sham TBS applied on the left side of the brain. In addition, subjects undergo the following:

" Pinch force: Subjects press a wedged instrument between the thumb and index finger as hard as they can during several trials every 10 seconds.

" Speed tapping: Subjects press a key on a computer keyboard as quickly as possible for 10 seconds, repeated for several trials.

" Simple reaction time: Subjects respond as quickly as possible to a "go" signal presented on a computer monitor by performing a quick wrist movement.

" Electromyography: Subjects' muscle activity is recorded using electrodes (small metal disks) filled with conductive gel and taped to the skin over the muscle.

Visits 2 and 3

Visit 2 is scheduled for one day after visit 1, and visit 3 is one week after visit 1. Participants do not have brain stimulation during these two visits, but they have TMS measurements, behavioral measurements, and electromyography (EMG) to see if the brain stimulation done during the first visit is still present after a period of time.

At all three visits, participants comp...

DETAILED DESCRIPTION:
OBJECTIVES:

Previous studies have demonstrated that single-pulse transcranial magnetic stimulation (TMS) applied to the primary motor cortex (MI) exerts a transient inhibitory effect on the contralateral MI. Furthermore, down-regulation of excitability in MI of one hemisphere by 1Hz rTMS results in increased excitability in the homologous MI accompanied by performance improvements in simple motor tasks performed by the hand ipsilateral to rTMS. It has been proposed that this phenomenon relies on interhemispheric disinhibition between both MI. Furthermore, interhemispheric disinhibition is also a promising method for boosting neurorehabilitation since interhemispheric disinhibition has been successfully applied in stroke patients to enhance motor cortex excitability and hand function or reduce aphasia. The purpose of this protocol is to test the hypothesis that interhemispheric disinhibition of the left MI by down-regulating activity in the right MI can be further enhanced by additional up-regulation targeting the left MI.

STUDY POPULATION:

We will study a total number of 72 healthy volunteers between the ages of 18-55.

DESIGN:

To test the hypothesis, subjects will be randomly allocated to one of 4 experimental sessions (parallel design). Subjects will receive different types of combined brain stimulation (1 Hz rTMS and Theta Burst Stimulation [TBS]) to the right and left MI. The primary outcome measure will be the amount of changes in cortical excitability, as reflected by recruitment curves (RC) of motor evoked potentials (MEPs) elicited by single-pulse TMS over the left MI. Additionally, we will test changes in short-interval intracortical inhibition (SICI) and facilitation (ICF) as well as the modulation of interhemispheric inhibition (IHI) between both MI. The secondary outcome measures will include simple motor tasks such as finger tapping, pinch force/acceleration and reaction time of the right hand.

In summary, we believe that this approach might identify additional effective strategies to enhance functional recovery after stroke and might provide deeper insight into the neural substrates involved in performance improvements after bilateral brain stimulation.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age between 18-55 years
  2. Able to perform tasks required by the study
  3. Willing and able to give consent

EXCLUSION CRITERIA:

Subjects are not eligible for this experiment if they:

1. Are unable to perform the tasks
2. Have history of severe alcohol or drug abuse, psychiatric illness
3. Have problems with movement of the hands
4. Are currently under medication with central acting drugs
5. Are left-handed
6. Have uncontrolled medical problems, such as heart, lung or kidney disease, epilepsy, or diabetes mellitus
7. Have a cardiac pacemaker, intracardiac lines, implanted medication pumps, neural stimulators, and metal in the cranium, with the exception of dental braces
8. Are pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72
Dates: Start 2006-11-03; Study Completion 2008-12-15

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Boroojerdi B, Battaglia F, Muellbacher W, Cohen LG. Mechanisms influencing stimulus-response properties of the human corticospinal system. Clin Neurophysiol. 2001 May;112(5):931-7. doi: 10.1016/s1388-2457(01)00523-5. PMID 11336911
- [Background] Chen R, Classen J, Gerloff C, Celnik P, Wassermann EM, Hallett M, Cohen LG. Depression of motor cortex excitability by low-frequency transcranial magnetic stimulation. Neurology. 1997 May;48(5):1398-403. doi: 10.1212/wnl.48.5.1398. PMID 9153480
- [Background] Di Lazzaro V, Oliviero A, Mazzone P, Pilato F, Saturno E, Dileone M, Insola A, Tonali PA, Rothwell JC. Short-term reduction of intracortical inhibition in the human motor cortex induced by repetitive transcranial magnetic stimulation. Exp Brain Res. 2002 Nov;147(1):108-13. doi: 10.1007/s00221-002-1223-5. Epub 2002 Sep 18. PMID 12373375